CLINICAL TRIAL: NCT01344252
Title: Topical Jelly and Intracameral Anesthesia Versus Subtenon Anesthesia, in Cataract Surgery: Preference and Surgical Conditions
Brief Title: Topical Jelly and Intracameral Anesthesia Versus Subtenon Anesthesia, in Cataract Surgery
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, Tomás Ortíz Basso, Ophthalmologist, Hospital Italiano de Buenos Aires
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1686
Record Dates: First submitted 2011-04-26; First posted 2011-04-29 (Estimated); Last update posted 2023-03-06 (Actual); Status verified 2015-03

CONDITIONS: Cataract Surgery Anesthesia
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Topical (Experimental)
  Interventions: Drug: Lidocaine
- subtenon (Active Comparator)
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — We will made anesthesia with topical lidocaine and compared with subtenon anesthesia

SUMMARY:
The options for anesthesia in cataract surgery described are: general, regional or local. The local strategy, it may be by periocular blocking(subtenon, peribulbar or retrobulbar), subconjunctival or topical. The risks faced by subconjunctival, peribulbar or retrobulbar, have made subtenon and topical strategies the most used. Likewise, to improve the effectiveness of the topical strategy was added gel topical lidocaine and intracameral dose of lidocaine.

Subtenon and topical anesthesia are two safe strategies and there were performed multiple studies showing that both are effective in controlling pain, but showing a slight superiority of subtenon. This difference does not appear to be clinically significant. In turn, the addition of gel and intracameral anesthesia, improved pain control. However, lack evidence to compare patient preference when using topical gel and intracameral anesthesia versus sub-Tenon anesthesia.

Multiple advantages has the topical anesthesia. Besides being a safe strategy for the patient, offers a rapid visual recovery, no generates blepharoptosis or diplopia postoperatively, subconjunctival hemorrhage and chemosis.

Because of this the investigators plan to conduct a study comparing the efficacy of gel topical and intracameral anesthesia versus subtenon anesthesia in cataract surgery with scleral incision, assessing the patient's preference Hypothesis: Topical administration of lidocaine in gel and intracameral anesthesia is a better strategy that subtenon anesthesia in cataract surgery

ELIGIBILITY:
Inclusion Criteria:

* bilateral cataract

Exclusion Criteria:

* refuse to participate, high surgical risk (ASA 4 or 5), allergy to lidocaine or other amide local anesthesics, inability to understand the informed consent, coagulation abnormalities, prior ophthalmologic surgery, small pupil, Fuchs dystrophy, lens luxation, uveitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-04

PRIMARY OUTCOMES:
number of subjects who prefer topical anesthesia. | 1 month
  The number of subjects who prefer topical anesthesia will measure at the end of the second surgery (1 month)

SECONDARY OUTCOMES:
intraoperative pain | 1 hour
  Amount of pain as verbal analog scale. Be evaluated at the end of surgery

CONTACTS AND LOCATIONS:
Locations (2):
- Argentina (2):
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Hospitalitaliano de buenos aires, CABA